CLINICAL TRIAL: NCT03479047
Title: Mechanical Ventilation Weaning Prediction Improved by Diaphragmatic Ultrasound Associated With the Rapid Shallow Breathing Index
Brief Title: Diaphragmatic Ultrasound Associated With RSBI Predict Weaning Issue: the Rapid Shallow Diaphragmatic Index (RSDI)
Acronym: CODEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2018-02
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Mechanical Ventilation; Mechanical Ventilator Weaning; Extubation; Diaphragm Ultrasound
Keywords: diaphragm ultrasound; spontaneous breathing trial; mechanical ventilation weaning; rapid shallow breathing index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventilated patients (Experimental): During a spontaneous breathing trial (SBT) we will simultaneously, for all included patient, assess diaphragmatic displacement (DD) using ultrasonography, respiratory rate (RR) and tidal volume (VT) on ventilator screen.
  Interventions: Diagnostic Test: assess diaphragmatic displacement (DD) using ultrasonography

INTERVENTIONS:
Diagnostic Test: assess diaphragmatic displacement (DD) using ultrasonography — During a spontaneous breathing trial (SBT) we will simultaneously, for all included patient, assess diaphragmatic displacement (DD) using ultrasonography, respiratory rate (RR) and tidal volume (VT) on ventilator screen.

SUMMARY:
The Rapid Shallow Breathing Index (RSBI) is the ratio between respiratory rate (RR) and tidal volume (VT). It is routinely used to predict mechanical ventilation weaning outcome in ICU patients. However RSBI doesn't reflect the muscular contribution of diaphragm or accessory muscles in generating tidal volume. Actually, diaphragmatic dysfunction can even delay weaning process, because accessory muscles are more fatigable than the diaphragm.

Hence, the investigators hypothesized that diaphragmatic displacement (DD) could be associated with RSBI in a new index named Rapid Shallow Diaphragmatic Index (RSDI) such as: RSDI = RSBI/DD.

The aim of this study is to compare the ability of the RSDI versus the traditional RSBI to predict weaning success in ready-to-wean patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mechanically ventilated patient > 24 hours
* Weaning ventilator phase (PEEP < 9 cmH2O and Support < 15 cm H2O)
* Ventilated via tracheostomy tube patient can be included on removal day of the cannula
* Patient's agreement to participate

Exclusion Criteria:

* Moribund patient
* Decision to forgo life sustaining therapy patient
* Patient with ventilation via tracheostomy tube before admission to ICU
* BMI > 45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Difference between the RSBI area and the RSDI AUC | 72 hours post-extubation
  Difference between the RSBI area under the receiving operator character curve (AUC) and the RSDI AUC in predicting success of mechanical ventilation weaning.

SECONDARY OUTCOMES:
Find a cut-off value for RSDI | 72 hours post-extubation
  - Find a cut-off value for RSDI with the best predicting accuracy for the weaning
Compare traditional RSBI values recorded with scientific publications | 72 hours post-extubation
Find reasons for non-extubation when criteria are gathered | 72 hours post-extubation
Estimate average duration of mechanical ventilation in central nervous system disorder patient | 72 hours post-extubation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spadaro S, Grasso S, Mauri T, Dalla Corte F, Alvisi V, Ragazzi R, Cricca V, Biondi G, Di Mussi R, Marangoni E, Volta CA. Can diaphragmatic ultrasonography performed during the T-tube trial predict weaning failure? The role of diaphragmatic rapid shallow breathing index. Crit Care. 2016 Sep 28;20(1):305. doi: 10.1186/s13054-016-1479-y. PMID 27677861
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] Farghaly S, Hasan AA. Diaphragm ultrasound as a new method to predict extubation outcome in mechanically ventilated patients. Aust Crit Care. 2017 Jan;30(1):37-43. doi: 10.1016/j.aucc.2016.03.004. Epub 2016 Apr 22. PMID 27112953
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Forgiarini LA Junior, Esquinas AM. The rapid shallow breathing index as a predictor of successful mechanical ventilation weaning: clinical utility when calculated from ventilator data. J Bras Pneumol. 2016 Jul-Aug;42(4):306. doi: 10.1590/S1806-37562016000000099. No abstract available. PMID 27832242